CLINICAL TRIAL: NCT03824717
Title: Minimum Effective Volume of 0.5% Ropivacaine for Ultrasound-Guided Infraclavicular Block
Brief Title: MEV 90 of 0.5% Ropivacaine In Infraclavicular Blocks
Acronym: MEV90ROPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112062
Record Dates: First submitted 2019-01-09; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Infraclavicular Brachial Plexus Block
Keywords: Ropivacaine; Brachial plexus block; Infraclavicular block

STUDY DESIGN:
Intervention Model Description: Biased coin design and up and down method to determine the minimum effective volume of Ropivacaine in ultrasound guided infraclavicular brachial plexus blocks.
Masking Description: There is no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine dosage (Other): Dose finding study - The volume of 0.5% ropivacaine used to achieve surgical anesthesia in infraclavicular brachial plexus block
  Interventions: Drug: Dose of ropivacaine

INTERVENTIONS:
Drug: Dose of ropivacaine — Biased coin design up and down dose finding study of 0.5% ropivacaine to achieve a successful infraclavicular brachial plexus block

SUMMARY:
Nerve blocks are routinely performed perioperatively to provide anesthesia and analgesia for various surgical procedures on the upper limb. These blocks are performed with the aid of an ultrasound machine to improve the success rate. Below the clavicle approach to these nerves is used for surgeries below the elbow, forearm and hand efficiently.

Ultrasound guidance for such blocks allows direct visualisation of the needle and the spread of the freezing medication (local anesthetic) in real-time therefore reducing complications and improving success rates of blocks. It may be possible that a smaller volume of local anesthetic in this setting may allow effective anesthesia while lowering the adverse effects. The aim of this study is to find out the lowest volume of the local anesthetic that will be effective in blocking the nerves adequately.

DETAILED DESCRIPTION:
This is a dose finding study. Volume assignment of ropivacaine will be carried out using a Biased Coin Design up and down method. In this method, the volume of local anesthetic (ropivacaine) administered to each patient will depends on the response of the previous patient. In the event of block failure, the next subject will receive an additional 2 mL of volume compared with the previous patient. In the event of block success, the next patient will receive either the same volume as the last patient or a 2 mL reduction in volume (per the biased coin design with a probability of the same volume being 0.9 and lower volume being 0.1). The first patient in the study will receive 30 mL and depending on the block success, the volume of the next block will be increased or decreased. The biased coin design is well described and established in other minimum volume studies.

All patients will have the block in the block room with standard monitoring (non-invasive blood pressure, pulse-oximetry, electrocardiogram) and mild sedation with midazolam and fentanyl. All blocks will be performed by staff anesthesiologists with a subspecialty in regional anesthesia and who work routinely in the block room or by a resident or fellow who is directly supervised by one of these staff anesthesiologist.

There will be two follow up telephone call to all patients enrolled in this study 24 hours post block insertion and one at 7 days to discuss length of block duration, any postoperative nausea/vomiting, any ongoing numbness or tingling, and overall satisfaction with the block. The participants will be informed of this phone call as part of the consent process and their telephone number will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years
* Amercian Society of Anesthesia physical status I, II, III
* Patients undergoing upper limb surgeries (with/without sedation)
* Ability to provide written informed consent

Exclusion Criteria:

* Patient refusal
* Known history of sensitivity or contraindications to study drugs
* Pregnant patients
* Infection at the site of administration of block
* Significant blood coagulation disorders
* Neurological deficits involving brachial plexus
* Patients on any medication which is known to have drug interactions with the study drugs
* Patients who receive general anesthesia/ narcotic supplements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
ED90 of 0.5% Ropivacaine | 30 minutes
  Volume used to achieve sensory and motor blockade (surgical anesthesia)

SECONDARY OUTCOMES:
Surgical anesthesia | 30 minutes
  Sensory and motor blockade tested using pin prick sensation ( 0 - normal sensation and can feel pin-prick, 1 - touch only, 2 - no sensation of touch or pinprick) and motor function of the ulnar, radial and median nerves.

OTHER OUTCOMES:
Duration of sensory anesthesia | 8 to 10 hours
  Duration of analgesia - time from administration of block to Visual analogue scale score more than 4 or patient request for first analgesic dose
Complications during block placement | 30 minutes
  Incidence of paresthesia during needle insertion, vascular or pleural puncture
Postoperative complications 24 hours and 7 days | 24 hours and 7 days
  Presence or absence of tingling, numbness, weakness of limb will be noted. Patient satisfaction as satisfied or unsatisfied will be noted.